CLINICAL TRIAL: NCT05967130
Title: Treatment of Chronic Relapsing Urinary Tract Infection With Bacteriophages in Renal Transplant Patients
Brief Title: Treatment Chronic UTI Post Kidney Transplant
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: drug not provided
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, nooshin dalili, Assistant Professor, Shahid Beheshti University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SBMU-
Record Dates: First submitted 2023-07-15; First posted 2023-08-01 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Urinary Tract Infections; Transplant-Related Disorder
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UC Positives (Experimental): Stable Transplanted Patients with Positive UC
  Interventions: Biological: Phage

INTERVENTIONS:
Biological: Phage — Inserting specific specimen of phages in to the bladder

SUMMARY:
Urinary tract infections (UTIs) with extended-spectrum -lactamase (ESBL)-positive Enterobacteriums (ESBL-E) are a common infectious complication of renal transplant recipients, with 10% of patients suffering from UTIs with ESBL-E within the first year posttransplant. Moreover, recurrence rates of UTI caused by ESBL-E are almost three times higher than those by cephalosporin-susceptible Enterobacteriums demonstrating the decreased efficacy of antibiotics in the treatment of these UTIs.

DETAILED DESCRIPTION:
According to each patient's urine culture, resistant urinary tract infections will be treated with specific phages and patients will be followed up with their urine cultures for response to therapy.

ELIGIBILITY:
Inclusion Criteria:

* Stable Kidney Transplant Recipients
* Stable Immunosupression Dose
* Stable Renal Function
* Resistant Urinary Infection with Positive UC

Exclusion Criteria:

* Rejection periods
* Frail Patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Urine culture | 1 week after administration
  Negative Urine Culture

CONTACTS AND LOCATIONS:
Overall Officials: Dalili, Principal Investigator — SBMU
Locations (1):
- Nooshin Dalili, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No